CLINICAL TRIAL: NCT06944145
Title: A Phase 2b Randomized, Single-Center, Double Blind, Placebo Controlled, 2-Arm Study to Investigate Orally Administered Combination Therapies (5-alpha Reductase Inhibitor + Raloxifene) Compared With Monotherapy (5-alpha Reductase Inhibitor + Placebo) in Adult Patients With Benign Prostatic Hyperplasia (BPH)
Brief Title: New Treatment Strategies and Epigenetic Biomarker for Management of Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aria F. Olumi, MD, Chief, Division of Urology, BIDMC, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000440; R01DK142211 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: BPH (Benign Prostatic Hyperplasia); Lower Urinary Track Symptoms
Keywords: BPH; SRD5A2; Finasteride; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Raloxifene Hydrochloride; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finasteride + Inactive Placebo Monotherapy (Active Comparator): Participants may be randomized into the Finasteride + Inactive Placebo Monotherapy arm.
  Interventions: Drug: Finasteride
- Finasteride + Raloxifene Combination Therapy (Experimental): Participants may be randomized into the Finasteride + Raloxifene Combination Therapy arm.
  Interventions: Drug: raloxifene; Drug: Finasteride

INTERVENTIONS:
Drug: raloxifene — Participants in the Finasteride + Raloxifene Combination Therapy Arm will receive both Finasteride and Raloxifene as their intervention.
  Participants randomized to the Finasteride + Raloxifene Combination Therapy arm will self-administer finasteride at 5 mg orally/day and raloxifene at 60 mg orally/day.
  Arms: Finasteride + Raloxifene Combination Therapy
Drug: Finasteride — Participants randomized to the Finasteride + Inactive Placebo Monotherapy arm will self-administer finasteride at 5 mg orally/day and placebo capsule daily.

SUMMARY:
SRD5A2 is a critical enzyme for prostatic development and growth, and the SRD5A2 inhibitor, finasteride, is used to treat benign prostatic hyperplasia (BPH). SRD5A2 is absent in 30% of normal adult men, which explains the resistance of a subset of patients to this commonly prescribed drug. This project proposes new combination therapies (5-ARI+raloxifene) and evaluates novel non-invasive biomarkers, based on alternative pathways that lead to prostatic enlargement.

DETAILED DESCRIPTION:
Over 90% of adult males develop lower urinary tract symptoms (LUTS) secondary to bladder outlet obstruction by age 80 secondary to benign prostatic hyperplasia (BPH). BPH, the most common proliferative abnormality in humans, negatively impact the quality of life of 210 million men globally, accounting for significant life years lost. This study proposes to clinically evaluate the mechanisms of resistance to 5α-reductase inhibitor, finasteride, one of the more common drugs used to manage BPH and associated LUTS. Ongoing work has focused on steroid 5α-reductase 2 (SRD5A2, aka: 5α-reductase 2 [5AR2]), the enzyme responsible for prostatic development and growth. Investigations have revealed that expression of SRD5A2 is variable, and in fact, 30% of men do not express SRD5A2 in prostate tissues. Previous work, shows that somatic suppression of SRD5A2 during adulthood is dependent on epigenetic changes associated with methylation of the promoter region of the SRD5A2 gene. Studies indicate that (1) methylation of the SRDA2 is regulated by direct binding of the DNA-methyl transferase 1 (DNMT1) protein to the SRD5A2 promoter; (2) the inflammatory mediators TNF-α, NF-kB, and IL-6 regulate DNMT1 binding and subsequent methylation of the SRD5A2 promoter region; (3) clinical conditions associated with increased inflammation, age, and obesity, are associated with decreased expression of SRD5A via epigenetic modification; (4) in the absence of prostatic SRD5A2, alternate estrogenic pathways are upregulated, leading to an androgenic-to-estrogenic switch in the prostate gland, thus creating alternate pathways for prostatic growth. Therefore, it is hypothesized that (1) non- invasive assessment of SRD5A2 methylation status in peripheral blood can be an excellent indicator for resistance to 5ARI therapy, and (2) in men demonstrating hypermethylation of SRD5A2 and low protein expression (patients suspected of being resistant to 5ARI therapy), combination therapy (Selective Estrogen Receptor Modulators [SERMs]+5ARI) will serve as a better treatment strategy. To demonstrate the clinical significance of epigenetic changes to SRD5A2 and confirm its role in regulating sensitivity to 5ARI treatment, and to examine the role of estrogenic signaling blockade, a clinical trial is proposed with: Specific Aim 1: To assess the role of combination therapy (5ARI + SERM) in the treatment of BPH and to determine whether methylation of SRD5A2 promoter is a predictor for response to therapy. Specific Aim 2: To prospectively evaluate whether non-invasive radiologic prostate inflammatory markers can predict circulating WBCs SRD5A2 promoter methylation.

ELIGIBILITY:
Inclusion criteria

1. ≥18 yrs old on the day of study consent;
2. Finasteride has been recommended for treatment of BPH by a physician;
3. PSA <20ng/ml within the last six months;
4. Willingness to maintain any current genitourinary medications (e.g., beta agonists, alpha blockers, anticholinergics);
5. Patient is able and willing to provide written informed consent.

Exclusion criteria

1. Active or past history of venous thromboembolism, including deep vein thrombosis, pulmonary embolism, and retinal vein thrombosis;
2. Previous diagnosis with any prostatic malignancy or precancerous lesions (atypical glandular foci);
3. History of pelvic radiation;
4. Actively receiving intravesical therapy for bladder cancer;
5. Received treatment with any demethylating medications (azacitidine, decitabine, zebularine, guadecitabine, hydralazine);
6. Current use of warfarin;
7. Prior treatment with 5ARI medications (e.g., Finasteride or Dutasteride) in the last year;
8. Diagnosed with diabetes mellitus;
9. Diagnosed with any neurodegenerative diseases;
10. History of allergic reaction to any intravenous (IV) iron replacement products;
11. Currently taking cholestyramine medication;
12. Contraindications to MRI examination, which may include:

    * Cardiac pacemaker
    * Intracranial clips, metal implants, or external clips within 10mm of the head
    * Previous metal injury in the eye or occupation risk to ferrous metal in the eye (e.g. metalworker)
    * Claustrophobia that cannot be managed with benzodiazepine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response to at 12 months after study enrollment | From enrollment to the end of treatment at 12 months
  The primary endpoint is the clinical response (yes-no) to therapy at 12 months after study enrollment between the combination and monotherapy treatment groups. Clinical response will be defined as ≥3-point increase in International Prostate Symptom Score between baseline and the 12-month timepoint, adjusting for baseline measure of International Prostate Symptom Score.
  The minimal International Prostate Symptom Score is 0, denoting no symptoms, and the maximum score is 35, denoting severe symptoms.

SECONDARY OUTCOMES:
Heterogeneity of clinical response to at 12 months after study enrollment by methylation score | From enrollment to the end of treatment at 12 months
  Assessing the clinical response (yes-no) to therapy at 12 months after study enrollment between the combination and monotherapy treatment groups. Clinical response will be defined as ≥3-point increase in International Prostate Symptom Score between baseline and the 12-month timepoint, adjusting for baseline measure of International Prostate Symptom Score. We will examine whether methylation score modifies the effect of treatment group on the primary endpoint by testing statistical interaction between treatment group and methylation score.
  The minimal International Prostate Symptom Score is 0, denoting no symptoms, and the maximum score is 35, denoting severe symptoms.
Comparison of mean International Prostate Symptom Score between study arms | From enrollment to the end of treatment at 12 months
  Mean 12-month International Prostate Symptom Score will be compared between study arms, adjusting for baseline International Prostate Symptom Score.
  The minimal International Prostate Symptom Score is 0, denoting no symptoms, and the maximum score is 35, denoting severe symptoms.
Comparison of mean International Index of Erectile Function Questionnaire scores between study arms | From enrollment to the end of treatment at 12 months
  Mean 12-month International Index of Erectile Function (IIEF) Questionnaire scores will be compared between study arms, adjusting for baseline International Index of Erectile Function score.
  A score of 0 to 5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The overall minimum score is 0, which indicates poor erectile function and the maximum score is 75 indicating good erectile function.
Correlation between methylation and MRI scores | From enrollment to the end of treatment at 12 months
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to the end of treatment at 12 months
  Comparison of treatment related adverse events by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Aria Olumi, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected throughout the trial. Data will be fully de-identified prior to sharing.
Supporting Information: ICF